CLINICAL TRIAL: NCT00046163
Title: A Phase IV, Multi-Center, Double-Blind, Parallel Group, Randomized, Placebo-Controlled Study to Assess the Clinical Benefit of Three Doses of Midodrine Hydrochloride (ProAmatine®) in Subjects With Neurogenic Orthostatic Hypotension
Brief Title: A Phase IV Study in Subjects With Neurogenic Orthostatic Hypotension
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated due to poor enrollment
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD 426-403
Record Dates: First submitted 2002-09-20; First posted 2002-09-23 (Estimated); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Hypotension, Orthostatic
Keywords: Neurology; Cardiology
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Midodrine

INTERVENTIONS:
Drug: midodrine hydrochloride (ProAmatine®)

SUMMARY:
We are seeking male and female patients to voluntarily take part in a clinical research study. Patients must be aged 18 or older and diagnosed with symptomatic orthostatic hypotension (low blood pressure while in the upright position) due to Parkinson's disease, multiple system atrophy, pure autonomic failure or autonomic neuropathies (i.e. neurogenic orthostatic hypotension). Symptoms of low blood pressure include dizziness, lightheadedness, changes in vision and generalized weakness upon standing. The main effect of the drug being studied is to increase blood pressure in the upright position so symptoms will decrease.

The purpose of this clinical study is to further assess the clinical effect of high dose midodrine hydrochloride (ProAmatine®), an approved treatment for orthostatic hypotension. During the course of the study, participants will receive either ProAmatine® or a placebo. Assessments will be made using questionnaires that measure symptom and activity levels. Blood pressure in the lying down, sitting and standing positions will be measured. Patients will also complete standing time assessments. They will be asked to remain standing without moving until they feel sufficiently lightheaded, or dizzy, or feel faint so that they would feel more comfortable sitting down.

ELIGIBILITY:
Inclusion Criteria:

* The male or female subjects must be 18 years of age or older and ambulatory. (Subjects must not require assistance with a walker or wheelchair to perform regular daily activities at all times.)
* Women of childbearing potential must have a negative serum beta HCG pregnancy test at screening and baseline.
* The subject has been diagnosed with symptomatic orthostatic hypotension due to Parkinson's disease, multiple system atrophy, pure autonomic failure or autonomic neuropathy (i.e. neurogenic orthostatic hypotension).
* The subject manifests one of the following symptoms while standing or has a history of one of the following when not treated for orthostatic hypotension: dizziness, lightheadedness, feeling faint or feeling like they may black out.
* The subject is willing and able to undergo the procedures required by this protocol including morning office visits, assessment completion, protocol compliance and participation in the wash-out period.
* The subject has signed an Institutional-Review-Board approved written informed consent form prior to any study procedures taking place.

Exclusion Criteria:

* The subject is a pregnant or lactating female.
* The subject has pre-existing sustained supine hypertension greater than 180 mm Hg systolic and 110 mm Hg diastolic.
* The subject is taking medications such as vasodilators, pressors, diuretics, ACE inhibitors, angiotensin receptor blockers, beta-blockers, combined alpha and beta-blockers, MAOI's, herbals or specific mixed effect medications.
* The Principal Investigator deems any laboratory test abnormality clinical significant.
* The subject has a diagnosis of any of the following disorders at the time of screening: pheochromocytoma; cardiac conditions including: congestive heart failure within the previous 6 months, myocardial infarction within the previous 6 months, symptomatic coronary artery disease, history of ventricular tachycardia, or uncontrolled cardiac arrhythmias; thyrotoxicosis; uncontrolled diabetes mellitus (uncontrolled defined as a HgbA1c greater than or equal to 10%); history of cerebrovascular accident, transient ischemic attack (TIA) or symptomatic carotid artery stenosis within the previous 6 months; history of coagulopathies; pulmonary hypertension; severe psychiatric disorders; renal failure (Creatinine equal to or greater than 2 times the upper limit of normal)
* The subject has a concurrent chronic or acute illness, disability, or other condition that might confound the results of the tests and/or measurements administered in this trial, or that might increase the risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-09-05 (Actual); Primary Completion 2003-08-06 (Actual); Study Completion 2003-08-06 (Actual)

PRIMARY OUTCOMES:
Average Standing Time | Visit 6, 1 hour post-dose
  Standing time was assessed after the participant and clinician questionnaires and blood pressure measurements are completed.
Average Standing Time | Visit 7, 1 hour post-dose
  Standing time was assessed after the participant and clinician questionnaires and blood pressure measurements are completed.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- United States (3):
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Neurological Associates of Delaware Valley, Upland, Pennsylvania
  - Diabetes & Glandular Disease Research Associates, PA,, San Antonio, Texas

REFERENCES:
- See also: The National Dysautonomia Research Foundation — http://www.ndrf.org
- See also: CenterWatch - Clinical Trials Resource Site — http://www.centerwatch.com